CLINICAL TRIAL: NCT01805544
Title: Satisfaction and Quality of Life in Patients With a Diagnosis of DVT (Deep Venous Thrombosis) Who Take Rivaroxaban
Brief Title: Satisfaction/Quality of Life With Rivaroxaban in DVT (Deep Venous Thrombosis) Indication
Acronym: SATORI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16409; XA1214FR (Other: Company internal)
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thrombosis
Keywords: SF36 questionnaire; Anti Clot Treatment Scale; Satisfaction; Quality of Life; Rivaroxaban; Prevention & control; Pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Personal Satisfaction; Pulmonary Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban: 20 mg po once daily, which is also the recommended maximum dose. SmPC recommendations are to be followed for renal impairment
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 20 mg po once daily, which is also the recommended maximum dose. SmPC recommendations are to be followed for renal impairment

SUMMARY:
National, multicenter, prospective, observational, non-interventional study. The objective is to determine if the switch from Vitamin K antagonists (VKA) to Xarelto in subjects treated with VKA with issues in deep venous thrombosis (DVT), and prevention of recurrent DVT and pulmonary embolism (PE) is associated with an improvement of the treatment satisfaction after 3 months. The treatment satisfaction will be measured by the Anti Clot Treatment Scale (ACTS) score.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject ≥ 18 years of age,
* With a diagnosis of acute DVT treated with VKA with issues for at least the 4 previous weeks (issues are assessed on medical judgment)
* Who intends to start rivaroxaban for treatment of deep vein thrombosis (DVT), and prevention of recurrent DVT and pulmonary embolism (PE) following an acute DVT
* With anticoagulation therapy planned for at least 3 months

Exclusion Criteria:

* Contra indication to the use of Xarelto as described in the Summary of Product Characteristics (SmPC); key contra indications are:

  * Hypersensitivity to the active substance or to any of the excipients listed in SmPC section 6.1.
  * Lesion or condition at significant risk of major bleeding
  * Concomitant treatment with any other anticoagulant agent
  * Clinically significant active bleeding
  * Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C
  * Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years old, with a diagnosis of acute DVT treated with VKA with issues, who switch from VKA to Xarelto
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change of the Anti Clot Treatment Scale (ACTS) score at 3 months compared with baseline score | After 3 months

SECONDARY OUTCOMES:
Change of ACTS score after 1 and 6 months of treatment | After 1 and 6 months
Continuation rate at 1, 3 and 6 months | After 1, 3 and 6 months
Change of SF36 score at 1, 3 and 6 months (health related quality of life determined by SF36 questionnaire) | After 1, 3 and 6 months
Physician's satisfaction at 1, 3 and 6 months assessed by a 5-point Likert scale response ("very satisfied", "satisfied", "neutral", "unsatisfied" or "very unsatisfied") | After 1, 3 and 6 months
Patient's compliance with VKA treatment at baseline and with Xarelto treatment at 1, 3 and 6 months assessed by the investigator as good (≥80%), average (50-80%) or poor (<50%) | After 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, France